CLINICAL TRIAL: NCT05339828
Title: Unroofing Curettage for Treating Simple and Complex Sacrococcygeal Pilonidal Disease
Brief Title: Unroofing Curettage for Pilonidal Disease
Status: Completed | Type: Observational
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: Pilonidal Disease surgery
Record Dates: First submitted 2022-02-26; First posted 2022-04-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pilonidal Disease; Recurrence; Healing Wound
Keywords: complex pilonidal disease; unroofing curettage; recurrence; Lay open technique
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unroofing curettage: Surgery was performed with the patient lying in the prone position under local anesthesia. Next, a local anesthetic agent comprising a solution of lidocaine (20 mg/mL) and adrenaline (0.0125 mg/mL) was diluted with distilled water in a 1:2 ratio and applied. The tract was identified by passing small artery forceps along its length and was then opened by cutting directly down onto the forceps. The sinus and all its tracts were completely unroofed, and the base was curetted to remove all necrotic content, hair, and granulation tissue using a dry gauze. The fibrotic back wall was left as intact as possible to avoid delayed healing.
  Interventions: Procedure: unroofing curettage

INTERVENTIONS:
Procedure: unroofing curettage — Surgery was performed with the patient lying in the prone position under local anesthesia. The tract was identified by passing small artery forceps along its length and was then opened by cutting directly down onto the forceps. The sinus and all its tracts were completely unroofed, and the base was curetted to remove all necrotic content, hair, and granulation tissue using a dry gauze. The fibrotic back wall was left as intact as possible to avoid delayed healing. Hemostasis was achieved using diathermy with no drainage needed.

SUMMARY:
This study aimed to investigate the outcomes of patients who underwent UC as the primary intervention for simple or complex SPD

DETAILED DESCRIPTION:
Sacrococcygeal pilonidal disease (SPD) is a well-known chronic inflammatory condition that affects young adults; There are many treatment options available today, from simple non-surgical methods to extensive flap procedures. However, elaborate treatment strategies can turn this easily treatable disease into a long-term surgical ordeal, causing complications worse than the primary disease itself.

While, UC is considered safe and effective for treating simple SPD, its suitability for treating complex disease is poor and controversial. To date, no studies have investigated the efficacy of UC specifically when treating complex SPD.

This is the first study to identify and compare efficacy and outcomes after UC in patients classified into simple and complex SPD groups.

This study was conducted at the Department of Surgery of the Diskapi Training and Research Hospital in Ankara, Turkey. The local ethics committee of the institution approved the study protocol (number 27/02, dated March 22, 2016), and written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18 years or older

Exclusion Criteria:

* acute pilonidal abscess
* poorly controlled
* diabetes mellitus,
* immunosuppressive or coagulation disorders,
* pregnancy and/or lactation,
* other acute surgical diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged 18 years or older who applied for simple and complex SPD treatment between April 2016 and September 2018 and preferred the UC surgery from all the treatment options offered by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Recurrence | 15 days
  After healing was complete, any new sinus orifice or discharge from the wound was defined as disease recurrence.

SECONDARY OUTCOMES:
complete healing time | 15 days
  time after surgery until the wound is completely epithelialized
VAS pain score | 15 days
  Visual analog scale for pain
time to return to daily activities | 15 days
  time after surgery until the to return to daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Engin Olcucuoglu, MD, Principal Investigator — Ankara Diskapi Training and Research Hospital
Locations (1):
- Ankara Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Nothing

REFERENCES:
- [Background] Kepenekci I, Demirkan A, Celasin H, Gecim IE. Unroofing and curettage for the treatment of acute and chronic pilonidal disease. World J Surg. 2010 Jan;34(1):153-7. doi: 10.1007/s00268-009-0245-6. PMID 19820992
- [Background] McCallum IJ, King PM, Bruce J. Healing by primary closure versus open healing after surgery for pilonidal sinus: systematic review and meta-analysis. BMJ. 2008 Apr 19;336(7649):868-71. doi: 10.1136/bmj.39517.808160.BE. Epub 2008 Apr 7. PMID 18390914
- [Background] Karakayali F, Karagulle E, Karabulut Z, Oksuz E, Moray G, Haberal M. Unroofing and marsupialization vs. rhomboid excision and Limberg flap in pilonidal disease: a prospective, randomized, clinical trial. Dis Colon Rectum. 2009 Mar;52(3):496-502. doi: 10.1007/DCR.0b013e31819a3ec0. PMID 19333052
- [Result] Olcucuoglu E, Sahin A. Unroofing curettage for treatment of simple and complex sacrococcygeal pilonidal disease. Ann Surg Treat Res. 2022 Oct;103(4):244-251. doi: 10.4174/astr.2022.103.4.244. Epub 2022 Oct 7. PMID 36304191